CLINICAL TRIAL: NCT01808690
Title: Effects of Metformin on Cardiovascular Function in Adolescents With Type 1 Diabetes
Brief Title: EMERALD: Effects of Metformin on Cardiovascular Function in Adolescents With Type 1 Diabetes
Acronym: EMERALD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Diabetes Association (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-1528; R56DK078645 (NIH)
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Results first posted 2020-02-05 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes
Keywords: Adolescent; Youth; Diabetes; Insulin Resistance; Cardiovascular; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Experimental): Metformin will be given at a dose of 1000 mg twice a day orally for three months to assess changes in insulin resistance compared to placebo.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo will be given at a dose of 1000 mg twice a day orally for three months to assess changes in insulin resistance compared to metformin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Diabetes is increasingly common among youth, forecasting early complications. Type 1 (T1D) cause early heart disease, shortening lifespan despite modern improvements in control of blood sugars and other risk factors for heart disease. Poor insulin action, otherwise known as insulin resistance (IR), is the main factor causing heart disease in type 2 diabetes (T2D), but the cause of increased heart disease in T1D is unclear. IR may contribute to heart disease in T1D as in T2D, as the investigators and others have found the presence of IR in T1D. Much less is known about IR in T1D, but a better understanding of its role in T1D is critical to understanding causes of heart disease in T1D. The investigators long-term goal is to understand the early causes of heart disease in diabetes so that we can prevent it. The investigators unique initial findings suggest that even reasonably well-controlled, normal weight, T1D youth are IR. The IR appears directly related to the heart, blood vessel, and exercise defects, but in a pattern that appears very different from T2D. The goals of this study are to determine the unique heart, blood vessel and insulin sensitivity abnormalities in T1D youth, and determine whether metformin improves these abnormalities. A clear understanding of these factors will help determine the causes, and what treatments could help each abnormality.

Hypothesis 1: Metformin will improve insulin function and mitochondrial function in T1D.

Hypothesis 2: Metformin will improve vascular and cardiac function in T1D.

All measures will be performed twice, before and after a 3-month randomized, placebo-controlled design where subjects are randomized to either metformin or placebo. The independent impact of insulin action as well as glucose levels, BMI, T1D duration, and gender on baseline outcomes and the impact of changes in insulin action, glucose levels and BMI on response to metformin will also be examined to help customize future strategies to prevent heart disease in T1D. This study will advance the field by providing new information about the role of poor insulin action in the heart disease of T1D, and whether improving insulin action in T1D is helpful. If a focus on directly improving insulin action in T1D youth is supported by our studies, the clinical approach to T1D management may significantly change.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents 12-21 years of age with type 1 diabetes (defined as having positive antibodies as well as insulin requirement)
2. Willing to consent for participation in study
3. Body Mass Index (BMI) >5% on growth charts

Exclusion Criteria:

1. Current use of medications known to affect insulin sensitivity: oral glucocorticoids within 10 days, atypical antipsychotics, immunosuppressant agents, metformin or thiazolidinediones.
2. Currently pregnant or breastfeeding women
3. Use of a thiazolidinedione within 12 weeks
4. Severe illness or Diabetic Ketoacidosis within 60 days
5. Macroalbuminuria
6. Hemoglobin A1c > 12%
7. Weight > 136.4 kg or < 42 kg, BMI < 5%
8. Creatinine > 1.2
9. Hemoglobin < 9
10. Major psychiatric or developmental disorder limiting informed consent
11. Implanted metal devices
12. Inability to tolerate ≥500mg twice a day of metformin

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 52 (Actual)
Dates: Start 2013-03; Primary Completion 2016-12-02 (Actual); Study Completion 2016-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Nadeau, MD, MS, Principal Investigator — University of Colorado/Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado and University of Colorado Denver Health Sciences Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tommerdahl KL, Baumgartner K, Schafer M, Bjornstad P, Melena I, Hegemann S, Baumgartner AD, Pyle L, Cree-Green M, Truong U, Browne L, Regensteiner JG, Reusch JEB, Nadeau KJ. Impact of Obesity on Measures of Cardiovascular and Kidney Health in Youth With Type 1 Diabetes as Compared With Youth With Type 2 Diabetes. Diabetes Care. 2021 Mar;44(3):795-803. doi: 10.2337/dc20-1879. Epub 2021 Jan 5. PMID 33402367
- [Derived] Bjornstad P, Schafer M, Truong U, Cree-Green M, Pyle L, Baumgartner A, Garcia Reyes Y, Maniatis A, Nayak S, Wadwa RP, Browne LP, Reusch JEB, Nadeau KJ. Metformin Improves Insulin Sensitivity and Vascular Health in Youth With Type 1 Diabetes Mellitus. Circulation. 2018 Dec 18;138(25):2895-2907. doi: 10.1161/CIRCULATIONAHA.118.035525. PMID 30566007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three (3) enrolled participants decided against participation in the study before randomization occurred.
Groups:
- Metformin: Metformin will be given at a dose of 1000 mg twice a day orally for three months to assess changes in insulin resistance compared to placebo.
  Metformin
- Placebo: Placebo will be given at a dose of 1000 mg twice a day orally for three months to assess changes in insulin resistance compared to metformin.
  Placebo
Period: Overall Study
Arm/Group | Metformin | Placebo
Started | 25 | 23
Completed | 24 | 21
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin | Placebo | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (2.3) | 15.9 (2.7) | 16.6 (2.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 24 | 22 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Insulin Sensitivity
Description: Hypothesis 1: Metformin will improve insulin function in Type 1 Diabetes. Insulin function will be measured using a euglycemic-hyperinsulinemic clamp procedure at both baseline and after 3 months of treatment. A clamp measures insulin sensitivity. A higher number indicates a better outcome; a lower number indicates a worse outcome.
Time Frame: Baseline, Month 3
Population: Metformin group: 1 participant lost to follow-up, 1 IV access problem Placebo group: 2 lost to follow-up, 2 IV access problems
Measure: Mean (Standard Deviation); unit: (mg/kg/min)/(insulin)
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 23 | 19
(mg/kg/min)/(insulin) | 12.2 (3.2) | -2.4 (3.6)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Insulin function was defined as M/I (mg/kg/min)/(insulin). Power calculations were based on data from a small study in youth with poorly controlled T1DM, which reported a significant increase in M/I in the 11 participants treated with Metformin. On the basis of the effect size reported in that study, a sample size of 25 per group and an alpha of 0.05 provided us with 93% power to detect a difference of 1 SD in the primary outcome of M/I; Test type: Superiority; p = 0.005, Regression, Linear — Threshold for statistical significance P=0.05; We also fitted multivariable models, which included sex, pubertal status, change in BMI, and baseline M/I

2. Secondary Outcome: Change in ADP Time Constant
Description: Hypothesis 1b: Metformin will improve mitochondrial function in Type 1 Diabetes. 31Phosphorus magnetic resonance spectroscopy (MRS) was used before, during, and after 90 seconds of near-maximal isometric exercise of the calf muscle for post-exercise muscle mitochondrial function. ADP time constant is the time for conversion of ADP → ATP and is a measure of muscle mitochondrial health (energy metabolism).
  A faster recovery is a better outcome; a slower recovery is a worse outcome.
Time Frame: Baseline, Month 3
Population: 22 participants had both pre/post MRS data
Measure: Median (Inter-Quartile Range); unit: seconds (s)
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 12 | 10
seconds (s) | 0.46 [-5.62 to 7.72] | -0.47 [-1.55 to 0.34]
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.46, Regression, Linear — Threshold for statistical significance P=0.05; Adjusted for the baseline value of the variable, sex, age, change in VO2peak, change in insulin sensitivity, and treatment condition

3. Secondary Outcome: Change in Pulse Wave Velocity (PWV)
Description: Hypothesis 2a: Metformin will improve central vascular function in Type 1 Diabetes via pulse wave velocity (PWV) by MRI. PWV is a measure of central arterial stiffness.
  A lower value indicates a better outcome.
Time Frame: Baseline, Month 3
Population: Number of participants analyzed differs from participant flow numbers because the institution's MRI scanner was unavailable during replacement.
Measure: Mean (Standard Deviation); unit: m/s
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 20 | 17
m/s | -1.1 (1.2) | 4.1 (1.6)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.04, Regression, Linear — Threshold for statistical significance P=0.05; We also fitted mutlivariable models, which included changed in SBP, change in BMI, and change in M/I

4. Secondary Outcome: Change in Central Arterial Intimal Medial Thickness (cIMT)
Description: Hypothesis 2a: Metformin will improve central vascular function in Type 1 Diabetes via central arterial intimal medial (cIMT) thickness by carotid ultrasound. cIMT is a measure used to diagnose the extent of carotid atherosclerotic vascular disease. The test measures the thickness of the inner two layers of the carotid artery-the intima and media.
  A lower result is a better outcome.
Time Frame: Baseline, Month 3
Population: Metformin: 1 lost to follow-up Placebo: 2 lost to follow-up
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 21
mm | -0.04 (0.01) | 0.00 (0.10)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.04, Regression, Linear — Threshold for significance P=0.05; We also fitted mutlivariable models, which included changed in systolic blood pressure, change in BMI, and change in M/I

5. Secondary Outcome: Change in Mitral Valve E/A Ratio by Echocardiogram
Description: Hypothesis 2b: Metformin will improve cardiac function in Type 1 Diabetes by echocardiogram.
  Mitral Valve E/A ratio is the ratio of early (E) to late (A) ventricular filling velocities.
  Ideal myocardial tissue relaxation is indicated by a ratio of >0.8 and <2.0.
Time Frame: Baseline, Month 3
Population: Metformin: 2 lost to follow-up Placebo: 2 lost to follow-up, 1 echocardiogram not performed
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 23 | 20
ratio | 1.55 (0.42) | 1.72 (0.34)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.01, Regression, Linear — Threshold for statistical significance P=0.05; Adjusted for the baseline value of BMI percentile, diabetes duration, and A1c

6. Secondary Outcome: Change in Aortic Wall Sheer Stress (WSS)
Description: Hypothesis 2a: Metformin will improve central vascular function in Type 1 Diabetes via Aortic Wall Sheer Stress (WSS) by MRI. WSS is a measure of central arterial stiffness.
  A lower value indicates a better outcome.
Time Frame: Baseline, Month 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: dyne/cm2
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 20 | 17
dyne/cm2 | -0.3 (0.4) | 1.5 (0.5)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.03, Regression, Linear — Threshold for statistical significance P=0.05; We also fitted mutlivariable models, which included changed in SBP, change in BMI, and change in M/I

7. Other Pre Specified Outcome: Change in Brachial Artery Distensibility
Description: Hypothesis 2a: Metformin will improve peripheral arterial stiffness in Type 1 Diabetes via Dynapulse.
  Peripheral arterial stiffness is measured by the distensibility of the arterial wall. Increased arterial stiffness results from reduced elasticity of the arterial wall.
  A higher result is a better outcome.
Time Frame: Baseline, Month 3
Population: Metformin: 1 lost to follow-up Placebo: 2 lost to follow-up
Measure: Mean (Standard Deviation); unit: %/mmHg
Arm/Group | Metformin | Placebo
Number analyzed (Participants) | 24 | 21
%/mmHg | 0.23 (0.19) | 0.16 (0.20)
Statistical Analysis 1: Comparison: Metformin vs Placebo; Test type: Superiority; p = 0.8, Regression, Linear — Threshold for significance P=0.05; [statistical method as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Metformin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23
Other Adverse Events (participants affected / at risk) | 10/25 | 2/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=25) | Placebo (N=23)
Gastrointestinal Side Effects (Gastrointestinal disorders) | 10 | 2 — nausea, diarrhea, reduced appetite, stomach pain

LIMITATIONS AND CAVEATS:
Results may not apply to prepubertal youth. Treatment duration limited to 3 months. MRI unavailable during scanner replacement. Lacked measure to monitor BGs during vascular assessments. Not all females studied in traditional follicular phase.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT01808690/Prot_SAP_000.pdf